CLINICAL TRIAL: NCT06181903
Title: The Effect of Emotional Freedom Technique Applied to Women With Risky Pregnancy on Mental Well-Being and Stress Level
Brief Title: The Effect of Emotional Freedom Technique on Mental Well-Being and Stress Level in Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra KARATAŞ OKYAY, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSUESRAKARATASOKYAY005
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Pregnant at Risk
Keywords: Pregnant; Well-being; Mental health; Stress; Emotional Freedom Technique
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional freedom technique group (Experimental): Emotional freedom technique will be applied to risky pregnant women in the emotional freedom technique group.
  Interventions: Behavioral: Emotional freedom technique group
- Control group (No Intervention): Pregnant women in the control group will not receive any intervention other than routine hospital care.

INTERVENTIONS:
Behavioral: Emotional freedom technique group — Control group
  Other Names: No Intervention
  Arms: Emotional freedom technique group

SUMMARY:
Emotional freedom technique will be applied to women with risky pregnancy. Emotional freedom technique group and control groups each consisted of 60 pregnant women.

DETAILED DESCRIPTION:
Objective In this experimental study, it was aimed to examine the effect of emotional freedom technique applied to women with risky pregnancy on mental well-being and stress levels.

Materials and Methods: This randomized controlled study will be conducted between February 2024 and August 2024 in Kahramanmaraş Necip Fazıl City Hospital Obstetrics and Gynecology Annex Building Obstetrics Outpatient Clinics with a total of 120 risk pregnant women (60 EFT, 60 control). EFT will be applied in the study. Women in the EFT group will receive EFT four times at one-week intervals. Pretest data will be obtained by filling out the Personal Information Form, Warwick-Edinburgh Mental Well-Being Scale (WEMWB), Prenatal Distress Scale - Revised Version before the Emotional Freedom Technique application. After the interventions, post-test data will be obtained by completing the Warwick-Edinburgh Mental Well-Being Scale (WEMWB), Prenatal Distress Scale - Revised Version. In addition, the Subjective Units of Experience (SUE) scale will be administered before and after each EFT intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Graduated from at least primary school
* Volunteering to participate in the research,
* Primiparous,
* Pregnant women who do not have conditions such as infection, wound, scar in the tapping areas.
* Pregnant women who meet any of the criteria in the Ministry of Health Risk Assessment Form for Pregnancy.

Exclusion Criteria:

* Pregnant women who participated in EFT or other antenatal classes/programs during the study period.
* Those who did not want to continue participating in the study,
* Those with a psychological problem according to the pregnant women's statements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of the level of Mental Well-Being | The Warwick-Edinburgh Mental Well-Being Scale will be administered to two groups of pregnant women on day one (first interview)
  The scale is a 14-item, self-report style scale. The scale consists of positive items including hedonic and eudaimonic dimensions of mental well-being, optimism, feeling useful, relaxation, interest in other people, being energetic and lively, coping with problems, clear thinking, feeling good, feeling close to other people, self-confidence, decision-making, love, interest in new things and being cheerful. The scale covers psychological well-being and subjective well-being and deals with the positive mental health of individuals. The scale is a five-point Likert scale with a minimum score of 14 and a maximum score of 70. Scoring of the scale is as follows: strongly disagree (1), disagree (2), somewhat agree (3), agree (4), strongly agree (5). All items of the scale are positive. High scores on the scale indicate high mental well-being.
Assessment of the level of Mental Well-Being | The Warwick-Edinburgh Mental Well-Being Scale will be administered to three groups of menopausal women at the last interview (after the 4th intervention at one week interval).
  The scale is a 14-item, self-report style scale. The scale consists of positive items including hedonic and eudaimonic dimensions of mental well-being, optimism, feeling useful, relaxation, interest in other people, being energetic and lively, coping with problems, clear thinking, feeling good, feeling close to other people, self-confidence, decision-making, love, interest in new things and being cheerful. The scale covers psychological well-being and subjective well-being and deals with the positive mental health of individuals. The scale is a five-point Likert scale with a minimum score of 14 and a maximum score of 70. Scoring of the scale is as follows: strongly disagree (1), disagree (2), somewhat agree (3), agree (4), strongly agree (5). All items of the scale are positive. High scores on the scale indicate high mental well-being.
Assessment of prenatal distress level | The Prenatal Distress Scale - Revised Version will be administered to two groups of pregnant women on day one (first interview)
  The scale determines pregnant women's social relationships, their physical and emotional symptoms during pregnancy, and their level of anxiety about themselves and their babies. The scale items have options ranging from "Not at all" (0), "A little" (1) and "Very much" (2), and the total score is obtained by summing the scores of the answers given to the scale items. A minimum score of 0 and a maximum score of 34 points are obtained from the scale. An increase in the total score obtained from the scale indicates an increase in the level of prenatal distress perceived by pregnant women.
Assessment of prenatal distress level | The Prenatal Distress Scale - Revised Version will be administered to three groups of menopausal women at the last interview (after the 4th intervention at one week interval).
  The scale determines pregnant women's social relationships, their physical and emotional symptoms during pregnancy, and their level of anxiety about themselves and their babies. The scale items have options ranging from "Not at all" (0), "A little" (1) and "Very much" (2), and the total score is obtained by summing the scores of the answers given to the scale items. A minimum score of 0 and a maximum score of 34 points are obtained from the scale. An increase in the total score obtained from the scale indicates an increase in the level of prenatal distress perceived by pregnant women.
Determining the level of anxiety | The Subjective Units of Experience (SUE) scale will be administered to two groups of pregnant women on day one (first interview)
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | One hour after the first interview, all pregnant women in all two groups will be administered the SUE (second measure)
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | Seven days after the first interview, all pregnant women in all two groups will be administered the SUE (third measurement)
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | One hour after the third measurement, all pregnant women in all two groups will be administered the SUE (fourth measurement)
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | Seven days after the fourth measurement, all pregnant women in all two groups will be administered the SUE (fifth measurement)
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | : One hour after the fifth measurement, all pregnant women in all two groups will be administered the SUE (sixth measurement)
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | Seven days after the sixth measurement, all pregnant women in all two groups will undergo the SUE (seventh measurement).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | One hour after the seventh measurement, all pregnant women in all two groups will be administered the SUE (eighth measurement)
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of pregnant women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Eda SEVER, Study Director — Kahramanmaras Sutcu Imam University; Esra GÜNEY, PhD, Study Director — Inonu University; Esra KARATAŞ OKYAY, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We don't share individual participant data with other researchers

REFERENCES:
- [Background] Irmak Vural P, Aslan E. Emotional freedom techniques and breathing awareness to reduce childbirth fear: A randomized controlled study. Complement Ther Clin Pract. 2019 May;35:224-231. doi: 10.1016/j.ctcp.2019.02.011. Epub 2019 Feb 15. PMID 31003663
- See also: Description citation link — https://pubmed.ncbi.nlm.nih.gov/31003663/